CLINICAL TRIAL: NCT01016561
Title: A Pilot Study of MR Imaging Based Intracavitary Brachytherapy for Cervical Cancer
Brief Title: Magnetic Resonance Imaging-Based Radiation Therapy and Cisplatin in Patients With Stage I, Stage II, Stage III, or Stage IV Cervical Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor accrual/enrollments
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 01809
Record Dates: First submitted 2009-11-18; First posted 2009-11-19 (Estimated); Results first posted 2021-05-05 (Actual); Last update posted 2021-05-05 (Actual); Status verified 2021-05

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Radiotherapy, Intensity-Modulated; Radiotherapy, Conformal; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm I (Experimental): Patients undergo external beam radiotherapy (3-dimensional conformal OR intensity-modulated) and 4-6 insertions of MRI-guided intracavitary brachytherapy over 8 weeks. Patients also receive cisplatin IV over 30-60 minutes for 5-6 weeks during radiotherapy.
  Interventions: Radiation: intracavitary balloon brachytherapy; Radiation: external beam radiation therapy; Radiation: intensity-modulated radiation therapy; Radiation: radiation therapy treatment planning/simulation; Radiation: 3-dimensional conformal radiation therapy; Drug: Cisplatin

INTERVENTIONS:
Radiation: intracavitary balloon brachytherapy
Radiation: external beam radiation therapy
  Other Names: EBRT
Radiation: intensity-modulated radiation therapy
  Other Names: IMRT
Radiation: radiation therapy treatment planning/simulation
Radiation: 3-dimensional conformal radiation therapy
  Other Names: 3D-CRT, conformal radiation therapy
Drug: Cisplatin

SUMMARY:
Rationale: Computer systems that allow doctors to create a 3 dimensional (3-D) picture of the tumor may help in planning radiation therapy and may result in more tumor cells being killed. Specialized radiation therapy that delivers a high dose of radiation directly to the tumor may kill more tumor cells and cause less damage to normal tissue. Drugs, such as cisplatin, may make tumor cells more sensitive to radiation therapy.

DETAILED DESCRIPTION:
PURPOSE: This clinical trial is studying magnetic resonance imaging-based radiation therapy and cisplatin in treating patients with stage I, stage II, stage III, or stage IV cervical cancer.Detailed DescriptionPRIMARY OBJECTIVES:

I. To evaluate the feasibility of using MRI based treatment planning for intracavitary brachytherapy treatment planning.

SECONDARY OBJECTIVES:

I. To evaluate the incidence of early toxicities, specifically genitourinary and gastrointestinal.

II. To evaluate the incidence of late toxicities, specifically genitourinary and gastrointestinal.

III. To evaluate local, regional, and distant recurrence rates. IV. To evaluate disease-free and overall survival rates. OUTLINE: Patients undergo external beam radiotherapy (3-dimensional conformal OR intensity-modulated) and 4-6 insertions of MRI-guided intracavitary brachytherapy over 8 weeks. Patients also receive cisplatin IV over 30-60 minutes for 5-6 weeks during radiotherapy.

After completion of study treatment, patients are followed at 6 weeks, every 4 months for 2 years, and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have histologically confirmed squamous cell, adenosquamous or adenocarcinoma of the cervix
* Subjects must have non-metastatic FIGO Stage Ia-IVa cervical cancer
* Claustrophobic subjects must agree to be sedated during MRI procedures
* ECOG performance status of 0-2

Exclusion Criteria:

* Subjects with an inability to tolerate MR imaging
* Subjects who have had prior surgery for treatment of disease other than exploratory laparotomy or biopsy
* Study subjects who have contraindication to MRI scanning such as but not limited to subjects with pacemakers, metal fragments in the eye or certain metallic implants
* Women of childbearing potential who have a positive result on screening serum pregnancy test

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-07; Primary Completion 2012-07 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Abramson Cancer Center of the Unviersity of Pennsylvania, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I: Patients undergo external beam radiotherapy (3-dimensional conformal OR intensity-modulated) and 4-6 insertions of MRI-guided intracavitary brachytherapy over 8 weeks. Patients also receive cisplatin IV over 30-60 minutes for 5-6 weeks during radiotherapy.
  intracavitary balloon brachytherapy
  external beam radiation therapy
  intensity-modulated radiation therapy
  radiation therapy treatment planning/simulation
  3-dimensional conformal radiation therapy
  Cisplatin
Period: Overall Study
Arm/Group | Arm I
Started | 0 (Despite all possible efforts to contact the PI/study team, no data are available to be reported)
Completed | 0 (Despite all possible efforts to contact the PI/study team, no data are available to be reported)
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Despite all possible efforts to contact the PI/study team members, no data are available to be reported
Arm/Group | Arm I
Number analyzed (Participants) | 0
Age, Categorical
Age, Continuous [unit: years]
Sex: Female, Male
Ethnicity (NIH/OMB)
Race (NIH/OMB)
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Using MRI for Intracavitary Brachytherapy Treatment Planning.
Description: Feasibility will be defined if no greater than 10% of patients experience one of the following events: a) patient is unable to tolerate 50% of MRI-based brachytherapy treatments and b) patient experiences any grade 4 acute ("early") non-hematologic toxicity attributed to brachytherapy. Acute toxicity occurs within 60 days of therapy.
Time Frame: Completion of study
Population: he study was terminated and the PI has left the institution. Despite all possible efforts to contact the PI/study team members, no data are available to be reported
Arm/Group | Arm I
Number analyzed (Participants) | 0

2. Secondary Outcome: Frequency of Grade 2 and Higher Gastrointestinal and Genitourinary Early Event Rates as Compared to Historical Series.
Time Frame: 60 days post treatment
Population: as for outcome 1
Arm/Group | Arm I
Number analyzed (Participants) | 0

3. Secondary Outcome: True Pelvis Failure
Time Frame: Time to local recurrence
Population: as for outcome 1
Arm/Group | Arm I
Number analyzed (Participants) | 0

4. Secondary Outcome: Pelvis Failure
Time Frame: Time to loco-regional recurrence
Population: as for outcome 1
Arm/Group | Arm I
Number analyzed (Participants) | 0

5. Secondary Outcome: Progression-free Survival
Time Frame: Time to recurrence
Population: as for outcome 1
Arm/Group | Arm I
Number analyzed (Participants) | 0

6. Secondary Outcome: Overall Survival
Time Frame: Time to death
Population: Not enough patients were accrued to the study for analysis.
Arm/Group | Arm I
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: The study was terminated and the PI has left the institution. Despite all possible efforts to contact the PI/study team members, no data are available to be reported
Arm/Group | Arm I
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes